CLINICAL TRIAL: NCT06724042
Title: First-in-human Phase 1a/b, Open-Label, Multicenter, Dose Escalation, Optimization and Expansion Study of ISM5939 in Patients With Advanced and/or Metastatic Solid Tumors
Brief Title: Study of ISM5939 in Patients With Advanced and/or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InSilico Medicine Hong Kong Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISM5939-101
Record Dates: First submitted 2024-12-01; First posted 2024-12-09 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Advanced and/or Metastatic Solid Tumors
Keywords: ISM5939; Ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1); ENPP1 inhibitor; Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Cisplatin; Docetaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Dose escalation (Experimental): An open-label dose escalation of ISM5939 administered orally as a single agent in patients with advanced or metastatic solid tumors.
  Interventions: Drug: ISM5939
- Part 2 Dose optimization (Experimental): ISM5939 will be administered orally as a single agent in patients with advanced or metastatic solid tumors in 2 selected dose levels to determine RP2D of ISM5939 monotherapy.
  Interventions: Drug: ISM5939
- Part 3 Dose expansion (Experimental): This will be an open-label evaluation of ISM5939 administered orally in combination with cisplatin, docetaxel, or pembrolizumab in patients with selected advanced solid tumors. Each of the combination cohort will start with safety run-in dose escalation for ISM5939. Subsequent subjects will then be enrolled in combination expansion cohorts with a fixed dose of ISM5939 selected by safety review committee.
  Interventions: Drug: ISM5939; Drug: Cisplatin; Drug: Docetaxel; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ISM5939 — ISM5939 tablets will be administered orally once daily (QD).
Drug: Cisplatin — Cisplatin will be administered intravenously in combination with ISM5939 on day 1 during each cycle.
  Arms: Part 3 Dose expansion
Drug: Docetaxel — Docetaxel will be administered intravenously in combination with ISM5939 on day 1 during each cycle.
  Arms: Part 3 Dose expansion
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously in combination with ISM5939 on day 1 during each cycle.
  Arms: Part 3 Dose expansion

SUMMARY:
This is a first-in-human Phase 1a/b, open-label, multicenter, dose escalation, optimization and expansion study of ISM5939 to evaluate the safety, tolerability, PK, PD, and preliminary antitumor activity of ISM5939 in patients with advanced or metastatic solid tumors.

The study will be conducted in 3 parts sequentially: Part 1 dose escalation ISM5939 monotherapy, Part 2 dose optimization to determine RP2D of ISM5939 monotherapy, and Part 3 dose expansion in 3 cohorts after initial safety run-in of ISM5939 combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years.
2. Patients with histologically or cytologically confirmed diagnosis of advanced/metastatic solid tumor that is either locally advanced and not amenable to curative therapy or stage 4 disease.
3. Patients must have tumor relapse/recurrence and be refractory to available SOC treatment, be intolerant to or ineligible for available SOC treatment, or have no SOC treatment available.
4. Patients enrolled in Part 3 (combination cohorts) must be acceptable and eligible for treatment with cisplatin, docetaxel, or pembrolizumab.
5. Measurable disease per RECIST version 1.1 or PCWG3 criteria for patients with metastatic castration-resistant prostate cancer.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1.
7. Patients must have recovered to Grade 1 or baseline levels from toxicity or AEs related to prior treatment for their cancer, excluding: Grade ≤2 neuropathy; alopecia of any grade, or skin pigmentation; Grade ≤2 hypothyroidism stable on hormone replacement therapy, Grade ≤2 anorexia or fatigue.
8. Patients must have an understanding, ability, and willingness to fully comply with study procedures and restrictions.
9. Patient must be capable of oral administration of ISM5939 and not have any clinically significant gastrointestinal abnormalities that may alter absorption.
10. Adequate bone marrow and organ function.
11. If receiving corticosteroids, patient must be maintained on a stable or decreasing dose for at least 7 days prior to Day 1.
12. Life expectancy ≥3 months in the opinion of the investigator.

Exclusion Criteria:

1. Patient has had prior systemic anti-cancer therapy within 3 weeks or at least 5 half-lives (whichever is shorter, but no less than 2 weeks) prior to Day 1.
2. Prior radiation therapy at the target lesion, unless there is evidence of disease progression and the prior radiation therapy is to have been completed at least 7 days before study drug.
3. Treatment with any investigational agent administered within 30 days or 5 half-lives, whichever is shorter, before the first dose of ISM5939.
4. Prior therapy with an ENPP1 inhibitor.
5. Currently receiving any of the CYP3A4/5 inhibitors/inducers, or CYP2C9 inhibitors, or inhibitors/inducers of MDR1, or medications known to prolong the QT interval that cannot be discontinued 14 days or 5 half-lives prior to Day 1.
6. Major surgery within 21 days prior to Day 1.
7. Patients with active (uncontrolled, metastatic) second malignancies or requiring therapy, or who have undergone potentially curative therapy with no evidence of the disease recurrence for at least 3 years prior to the first dose of study treatment.
8. Patients with a primary CNS tumor.
9. Patient has uncontrolled hypertension, or heart disease and/or cardiac repolarization abnormality, or uncontrolled systemic infection.
10. Other medical illness that, in the opinion of the investigator, may impact the safety of the patient or the objectives of the study.

Other protocol inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) occurrence | Day 1 up to Day 28 for Part 1 and Day 1 up to Day 21 for Part 3 safety run-in dose escalation period
  DLT is defined as any of the adverse event which meets DLT criteria if assessed at least possibly related to study treatment and not clearly related to progressive disease or other extraneous cause and occurring during the DLT period.
Adverse events (AEs) | Approximately 36 months
  Incidence and severity of AEs will be evaluated based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 [NCI CTCAE v5.0]).
Recommended Phase 2 doses (RP2Ds) | Approximately 36 months
  The maximum tolerated dose (MTD) or RP2Ds in patients with advanced or metastatic solid tumors will be determined based on the available data of safety and tolerability, PK, PD and preliminary activity from all dosed patients.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Approximately 36 months
  Blood samples for Pharmacokinetics (PK) analysis will be assessed after dose of ISM5939.
Area under the concentration-time curve (AUC) | Approximately 36 months
  Blood samples for Pharmacokinetics (PK) analysis will be assessed after dose of ISM5939.
Terminal half-life (t1/2) | Approximately 36 months
  Blood samples for Pharmacokinetics (PK) analysis will be assessed after dose of ISM5939.
Objective response rate (ORR) | Approximately 36 months
  ORR is defined as the percentage of participants with Complete Response or Partial Response.
Duration of response (DOR) | Approximately 36 months
  DOR is defined as the time from the first tumor assessment when the Complete Response/Partial Response is met to the date of disease progression or death, which occurs first.
Disease control rate (DCR) | Approximately 36 months
  DCR is defined as the percentage of participants with Complete Response or Partial Response or Stable Disease (persisted for at least 6 weeks).
Best overall response (BOR) | Approximately 36 months
  BOR is defined as the best response from the initial oral dose of ISM5939 until disease progression, initiation of another anti-tumor treatment, or early withdrawal (whichever occurs first). Confirmation of CR and PR is required.